CLINICAL TRIAL: NCT07254559
Title: Integrated Physiomarker, Biomarker and Clinical Predictive Analytics for Early Warning of Sepsis and Necrotizing Enterocolitis in Very Low Birth Weight Infants: Pilot Randomized Clinical Trial to Test Feasibility of Integrated Predictive Monitoring for Sepsis and NEC
Brief Title: Integrated Predictive Monitoring for Sepsis and Necrotizing Enterocolitis
Acronym: PREMO (K)
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Brynne Sullivan, Associate Professor of Pediatrics, University of Virginia
Other Study IDs: 21237; K23HD097254 (NIH); IER 231718 (Other: US NIH)
Record Dates: First submitted 2025-11-03; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Necrotising Enterocolitis Neonatal
MeSH Terms: conditions — Sepsis; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
Behind the scenes pilot trial in the computer lab involving chart review to use neonatal intensive care unit data to create computer models predicting sepsis and necrotizing enterocolitis in very small premature infants

ELIGIBILITY:
Inclusion Criteria:

* Less than 1500 grams at birth

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonatal intensive care patients of very low birth weight (VLBW) (<1500g)
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Presence of sepsis or necrotizing enterocolitis | Before end of NICU stay
  binary

CONTACTS AND LOCATIONS:
Overall Officials: Brynne Sullivan, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT07254559/Prot_SAP_000.pdf